CLINICAL TRIAL: NCT00489658
Title: Efficacy and Safety of an Eflornithine + Nifurtimox Combination for Treatment of Late-Stage Human African Trypanosomiasis (HAT) in West Nile, Uganda
Brief Title: Eflornithine + Nifurtimox Late-Stage Human African Trypanosomiasis (HAT)in West Nile, Uganda
Acronym: NECS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Because of unexpectedly reduced disease prevalence in the study area, a pragmatic decision was taken to terminate recruitment in March 2003.
Sponsor: Epicentre (Other)
Collaborators: Médecins Sans Frontières, France (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NECS
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Trypanosomiasis, African
Keywords: Human African trypanosomiasis; sleeping sickness; Trypanosoma brucei gambiense; combination; eflornithine; nifurtimox; Human African trypanosomiasis (sleeping sickness) due to Trypanosoma brucei gambiense in the late stage (stage 2 or meningo-encephalitic)
MeSH Terms: conditions — Trypanosomiasis, African | interventions — Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Eflornithine plus Nifurtimox combination therapy

SUMMARY:
This case series study follows on a terminated randomised clinical trial in a nearby location of Uganda, in which the combination of eflornithine + nifurtimox showed very promising efficacy and safety. The study's purpose is to evaluate the efficacy and safety of this combination in a larger group of late-stage Human African trypanosomiasis (sleeping sickness) patients.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2 infection with Trypanosoma brucei gambiense diagnosed within the previous 14 days, as defined by either of the following: (i) Presence of trypanosomes in blood or lymph node fluid and WBC count in CSF > 5 / mm3, or (ii) Presence of trypanosomes in the CSF with any CSF WBC count
* Residence in the study area
* Written informed consent (to be obtained from parent/guardian for children under 18 years and patients with impaired cognition)

Exclusion Criteria:

* Pregnancy or clinical history suggestive thereof
* Weight < 10 Kg
* History of any HAT treatment within the previous 24 months
* Inability to undergo hospitalisation or attend follow-up visits during the 24 months following discharge
* Severe anemia (Hb< 5g/dl)
* Active tuberculosis (sputum positive)
* HIV positive (if patient has been tested and results are known)
* Severe renal or hepatic failure
* Bacterial or cryptococcal meningitis
* Other severe underlying diseases upon admission
* Refugee status

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-10

PRIMARY OUTCOMES:
Treatment failure (death within 30 days of inclusion, or later if judged as related to Human African trypanosomiasis; termination of treatment due to adverse events; evidence of infection relapse at or after discharge, up to 24 months post discharge) | 24 months

SECONDARY OUTCOMES:
Occurrence and severity of serious clinically apparent adverse events | treatment period and up to one month post discharge
Occurrence and severity of biochemical (ALAT, creatinine, bilirubin) and haematological (abnormal total and differential leukocyte count, haemoglobin) adverse events | treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Piola, MD MSc, Principal Investigator — Epicentre; Gerardo Priotto, MD MPH, Study Director — Epicentre
Locations (1):
- Yumbe District Hospital, Yumbe, Yumbe District, Uganda

REFERENCES:
- [Background] Priotto G, Fogg C, Balasegaram M, Erphas O, Louga A, Checchi F, Ghabri S, Piola P. Three drug combinations for late-stage Trypanosoma brucei gambiense sleeping sickness: a randomized clinical trial in Uganda. PLoS Clin Trials. 2006 Dec 8;1(8):e39. doi: 10.1371/journal.pctr.0010039. PMID 17160135